CLINICAL TRIAL: NCT05937945
Title: Uncovering Osteoporosis Clinical Trials: Firsthand Patient Insights Into Clinical Trial Experiences
Brief Title: Studying Patient Experiences in Osteoporosis Clinical Trials
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 83312301
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Osteoporosis
Keywords: osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical trials for osteoporosis are designed to assess the safety and effectiveness of novel osteoporosis treatments. These trials play a crucial role in establishing whether these new treatments outperform existing options and provide substantial evidence to support their adoption within the wider population.

The primary aim of this particular study is to investigate the experiences of individuals diagnosed with osteoporosis who participate in a distinct clinical trial involving a medical intervention. The focus will be on closely monitoring the rates of trial completion and withdrawal among these participants.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with osteoporosis
* Patient has self-identified as planning to enroll in an observational clinical trial
* Patient is a minimum of 18 years or older

Exclusion Criteria:

* Pregnant or nursing patients
* Inability to perform regular electronic reporting
* Patient does not understand, sign, and return consent form

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Osteoporosis patients who are actively considering enrolling in an observational clinical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to join in an osteoporosis clinical trial | 3 months
Rate of patients who remain in osteoporosis clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu C, Liu N, Xia Y, Zhao Z, Xiao T, Li H. Osteoporosis and sarcopenia-related traits: A bi-directional Mendelian randomization study. Front Endocrinol (Lausanne). 2022 Sep 14;13:975647. doi: 10.3389/fendo.2022.975647. eCollection 2022. PMID 36187130
- [Background] Bell A, Kendler DL, Khan AA, Shapiro C M M, Morisset A, Leung JP, Reiner M, Colgan SM, Slatkovska L, Packalen M. A retrospective observational study of osteoporosis management after a fragility fracture in primary care. Arch Osteoporos. 2022 May 6;17(1):75. doi: 10.1007/s11657-022-01110-z. PMID 35513573
- [Background] Amer M, Noor S, Kashif SM, Nazir SUR, Ghazanfar T, Yousaf S. Evaluation of Disease Related Knowledge in Patients of Osteoporosis: An Observational Study. Altern Ther Health Med. 2021 Jun;27(S1):97-103. PMID 32663187

DOCUMENTS (1):
  • Informed Consent Form (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/45/NCT05937945/ICF_000.pdf